CLINICAL TRIAL: NCT03872895
Title: Adjustment of Adopted Adolescents in Their Families
Acronym: EEAA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Catholic University, Italy (Other); University of Oslo (Other); University of Seville, Spain (Unknown)
Responsible Party: Sponsor
Other Study IDs: D18-PO16
Record Dates: First submitted 2019-01-25; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-01

CONDITIONS: Adoption; Adolescent Behavior; Family Relations
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The adjustment of adopted adolescents has been studied in the U.S. and England, but few other European countries have conducted research into this topic. As countries differ greatly in their cultural practices, a comparative study of the adjustment of internationally adopted teenagers in 4 European countries (France, Italy, Spain, Norway) is planned. The adjustment of teens and their families will be studied in relation to the openness of communication related to adoption within the families.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the status of internationally adopted adolescents in relation to the characteristics of their families, and to explore the similarities and differences in 4 different European countries. Parents and adolescents will complete questionnaires which incorporate and adapt many standard measures. The parent questionnaire includes components of : a) Family Adjustment and Cohesion Scale (FACES), b) Strengths and Difficulties Questionnaire for parents (SDQ-parent), c) Parent Stress Index (PSI), d) Adoption Satisfaction Questionnaire (ASQ), d) Brodzinsky Scale (openness in family communication related to adoption), and e) basic demographic information.

The adolescent questionnaire includes elements of : a) SDQ-adolescent, b) Health Behavior in School Children questionnaire (HBSC), c) Life Orientation Test-Revised (LOT-R), d) Lee Scale (Discrimination Scale for Adoptees).

It is hoped that the study will permit a better understanding of the experiences of families and their children after international adoption. This knowledge will help potential adoptive families as well as families who have already adopted. This information is not yet available in a European context. In addition, the information will be valuable to adoption professionals. Moreover, the opportunity to compare outcomes and experiences of families and adolescents in 4 European countries will allow a better understanding of the contribution of different cultural contexts to these outcomes. It is hypothesized that different cultural practices and beliefs about adoption likely impact the experience of adoption by adolescents and parents. A better understanding of this dynamic will be useful clinically as well as at the community level and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Parents: have an internationally adopted adolescent between ages of 11-17 years child arrived in the family at least 6 months ago Adolescents: internationally adopted, between ages of 11-17 years arrived in the family at least 6 months ago

Exclusion Criteria:

* Parents: unwilling or unable to complete questionnaire Adolescent: unwilling or unable to complete questionnaire

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents who have an internationally adopted adolescent between ages of 11-17 years, and whose child arrived in the family at least 6 months ago, as well as internationally adopted adolescents between ages of 11-17 years who arrived in the family at least 6 months ago
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Openness of family communication related to adoption (standardized scale developed by David Brodzinsky) | past 30 days
  Openness to family communication about the subject of adoption will be assessed using the Brodzinsky standardized scale. This will be correlated to adolescent outcomes (adjustment to family, school, and community) using constructed variables drawn from the Health Behavior in School Children questionnaire

SECONDARY OUTCOMES:
Parent Stress (using PSI, Parent Stress Index) | past year
  Parent Stress will be measured using the widely-used Parent Stress Index. This scale contains 36 items which are completed by parent self-report. The items are combined to form a Total Stress scale. Scoring results in a percentile profile. The normal range=15th-80th percentile. Scores at or above the 85th percentile are considered high (more stress) and Defensive Reponding scores at 10 or below are considered extremely low. Cronbach's alpha for internal consistency: minimum =0.8, max=.91, and average=.85. This scale (first published in 1990 by Abdin) has been used and cited in over 4900 scientific papers.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Miller, MD, Study Chair — GHU Ste Anne
Locations (1):
- Hospital SAINTE ANNE, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided